CLINICAL TRIAL: NCT05992389
Title: Evidence Driven Indoor Air Quality Improvement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospital Srebrnjak (Other)
Responsible Party: Principal Investigator, Mirjana Turkalj, MD, Professor, MD, PhD, Children's Hospital Srebrnjak
Other Study IDs: SCH-EU101057497
Record Dates: First submitted 2023-05-12; First posted 2023-08-15 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Asthma in Children; Pollution; Exposure
Keywords: indoor air quality; asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with asthma: School aged participants (6-14 yrs) with an established diagnosis of asthma
- Non-asthmatic subjects (healthy control): School aged participants (6-14 yrs), non-asthmatic subjects (negative history of allergic diseases)

SUMMARY:
The aim is to identify the underlying disease mechanisms driving specific asthma phenotypes as well as certain disease outcomes and their relation to impaired indoor air quality. This may also help in underpinning specific target mechanisms in order to personalize and improve current treatment options in childhood asthma and develop more successful prevention strategies. This will be done by combining data from detailed clinical phenotyping with multiple -omics data.

DETAILED DESCRIPTION:
A recent report from the European Environmental Agency (EEA) shows that as many as 417 000 deaths per year in large European cities are caused by long-term exposure to air pollution (EEA 2018). Children are more sensitive to environmental risks than adults. Environmental pollution (impaired air quality) has been linked to asthma development. Asthma is the most common chronic disease in children, with estimations that one in every five children will develop asthma during childhood. The effects of poor air quality most likely act synergistically with other predisposing and environmental factors, and in a cumulative manner. Additionally, asthma in children is considered to be a complex syndrome encompassing a number of different disease subtypes (phenotypes) driven by distinct yet discrete underlying pathophysiological mechanisms (endotypes). Detailed characterization of these pheno- and endotypes in asthma, as well as disease and treatment outcomes resulting from them still remain elusive.

The modern way of life, especially in the light of the COVID-19 ('CO' stands for corona, 'VI' for virus, 'D' for disease, and '19' for 2019 (year first identified)) pandemic, implies that people spend up to 90% of our time indoors. Certain studies suggest that indoor air quality may be significantly worse than outdoors and the regulation of indoor air quality falls much behind the legislative and guidelines in outdoor air quality. It is reasonable to believe that indoor air quality affects human health (risk for allergy, asthma, and specific disease subtypes) at least as much as outdoor pollutants, if not more.

For the Evidence Driven Indoor Air Quality Improvement Srebrnjak Children's Hospital (EDIAQI SCH 2021) cohort, 200 school aged children (6-14 years) from the Croatian capital and its surroundings (Zagreb) will be recruited to this study from the outpatient clinic at the Srebrnjak Children's Hospital (SCH) in Zagreb, Croatia, which is the national Referral Centre of the Croatian Ministry of Health for Clinical Allergology in children.

150 of them with the diagnosed asthma and 50 participants their matching control, non-asthmatic subjects.

Following an expert (physician, experienced allergy/pulmonology specialist) confirmed diagnosis of asthma and after obtaining an informed consent from the children's caregivers/children themselves (according to local legislative), participants undergo a standard battery of diagnostic tests, examinations and procedures as a part of their routine asthma management plan. This study will also involve clinical follow-up visits (approximately every 3-6 months, according to Global Initiative for Asthma (GINA) guidelines). As a part of this research, certain biological samples (blood, exhaled breath condensate, induced sputum) will be collected both at baseline and follow-up visits, aiming at using biological samples left over from routine diagnostics whenever possible and using minimally invasive methods at all times.

The study will include visits:

1. Initial (screening) visit (First patient first visit- V0 +3 months): written consent, assessment of inclusion and exclusion criteria, physical examination, anthropometric measurements, skin prick test (SPT), Specific Immunoglobulin E (sIgE) (+ISAC), Atopy patch test (APT), spirometry, fractional exhaled nitric oxide (FENO), questionnaires, blood sampling, buccal cells swabs, exhaled breath condensate (EBC), induced sputum
2. First follow-up visit- V1 (V0 + 3-6 months): questionnaires, spirometry, FENO, anthropometric measurements, asthma control assessment
3. Second follow-up visit- V2 (V0 + 6-12 months): questionnaires, spirometry, FENO, anthropometric measurements, asthma control assessment
4. Third follow-up visit- V3 (V0 + 9-18 - months): questionnaires, spirometry, FENO, anthropometric measurements, asthma control assessment
5. Fourth follow-up visit (V0 + 21 months): questionnaires, spirometry, FENO, anthropometric measurements, asthma control assessment
6. Last visit (last patient last visit- V0 + 24 months): anthropometric measurements, SPT, sIgE (+ISAC), APT, spirometry, FENO, questionnaires, blood sampling, buccal cells swabs, EBC, induced sputum, asthma control assessment, final assessment of the study outcome measures, check and document consumption, adherence, preventive measures.

ELIGIBILITY:
Inclusion Criteria:

* school aged participants with asthma (patients with a clinical diagnosis of asthma (according to European Respiratory Society (ERS) and American Thoracic Society (ATS) guidelines) for at least a year , being on a stable dose of anti-inflammatory treatment for at least one month with partially controlled or uncontrolled asthma according to GINA guidelines)
* non-asthmatic school aged participants (matching control subjects)
* signed informed consent, .
* additional inclusion criteria include clinically significant allergy to indoor and outdoor allergens, with positive skin prick test (SPT) and specific IgE levels (>0.7 kUA/L) (UA = allergen-specific unit)

Exclusion Criteria:

* known inborn or perinatal pulmonary disease;
* pulmonary malformation;
* oxygen therapy after birth with a duration of more than 24h;
* ventilator support or mechanical ventilation after birth;
* diagnosis of cystic fibrosis;
* primary ciliary dyskinesia;
* heart failure diagnosed after birth affecting pulmonary circulation;
* major respiratory diseases such as e.g. interstitial lung disease,
* acute respiratory infection at recruitment,
* use of systemic corticosteroids,
* recent asthma-related visit to emergency department (in the past three weeks)
* coexistence of other serious chronic illness. Moreover, children will be excluded from study visits and biomaterial collection in the case of fever of at least 38.5°C during the last two weeks prior to the planned visit.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Total of 200 children will be recruited for this study. 150 school aged children with asthma (6-14 years) from the Croatian capital and its surroundings (Zagreb) will be recruited to this study. These participants will be recruited from the outpatient clinic at the Srebrnjak Children's Hospital in Zagreb, Croatia, as well as matching control participants (non-asthmatic subjects, N=50).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in the number of asthma exacerbations and severity | 6 months
  The exacerbation rate and exacerbation severity will be recorded along with the treatment use (reliever medication, use of oral and parenteral corticosteroids etc.) During the patient examination the questionnaire will be used to record the number of asthma exacerbations and the therapy used.
  Asthmatic patients will be regularly controlled even more often in case of exacerbations.

SECONDARY OUTCOMES:
Change of asthma control | 6 months
  Childhood Asthma Control Test (C-ACT) questionnaire will be used to tell us if the asthma treatment plan is optimal and if asthma is being properly controlled. For children 4 to 11 years maximal score is 27, and for those older then 12 years maximal score is 25. Higher scores reflect greater asthma control, and if the score is 19 or less may be a sign that asthma is not controlled as well as it could be.
  Asthmatic patients will be regularly controlled even more often in case of exacerbations.
Lung function tests | 6 months
  Forced expiratory volume in one second (FEV1), Forced vital capacity (FVC) and the ratio of the two volumes (FEV1/FVC) will be recorded for each patient at each visit. Both FEV1 and FVC are measured in liters
  FEV1 is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, measured in liters.
  Asthmatic patients will be regularly controlled even more often in case of exacerbations.
Fractional exhaled nitric oxide (FeNO) | 6 months
  FeNO test measures the level of nitric oxide gas in an exhaled sample of breath. It is measured in "parts per billion" (ppb).
  Asthmatic patients will be regularly controlled even more often in case of exacerbations.
Use of controller medication | 6 months
  Type and dose of controller medication wil be monitored and recorded. Asthmatic patients will be regularly controlled even more often in case of exacerbations.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Srebrnjak, Zagreb, Croatia